CLINICAL TRIAL: NCT04780737
Title: Prophylactic Cholecystectomy is Not Mandatory in Patients Candidate to the Resection for Small Intestine Neuroendocrine Neoplasms: a Propensity Score-matched and Cost-minimization Analysis
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Carlo Ingaldi, MD, Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: RAC 164/2017/ O/Oss
Record Dates: First submitted 2021-01-08; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Neuroendocrine Tumors; Surgery; Gut Tumor
MeSH Terms: conditions — Neuroendocrine Tumors; Digestive System Neoplasms | interventions — Cholecystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prophylactic cholecystectomy: Patient who undergo resection of primary ileal neuroendocrine tumor and contemporarly cholecystectomy
  Interventions: Procedure: Cholecystectomy
- On-demand cholecystectomy: Patient resected for primary ileal neuroendocrine tumor, treated with cholecystectomy in a different operation and only if needed, for the development of biliary stone disease
  Interventions: Procedure: Cholecystectomy

INTERVENTIONS:
Procedure: Cholecystectomy — Laparoscopic or laparotomic cholecystectomy

SUMMARY:
To evaluate two competitive strategies in patients undergoing resection of Small-intestine Neuroendocrine neoplasms (Si-NEN): Prophylactic Cholecystectomy (PC) versus On-demand delayed cholecystectomy

DETAILED DESCRIPTION:
This is a retrospective study based on 230 Si-NENs candidates to the primary tumor resection. Patients were divided into two arms: PC and OC. Propensity score matching was performed, reporting the d value. The primary outcome was the re-hospitalization rate for any cause. The secondary endpoints were the re-hospitalization rate for biliary stone disease (BSD), the mean number of re-hospitalization (any cause and BSD), the complication rate (all and severe), and the total costs. A P-value < 0.05 was considered significant, and NNT< 10 was considered clinically relevant.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of Si-NEN;
* resection of the primary tumor with or without concomitant cholecystectomy;
* absence of a history of a biliary stone disease or cholecystectomy before Si-NEN diagnosis

Exclusion Criteria:

- presence of a history of a biliary stone disease or cholecystectomy before Si-NEN diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For each patient sex, age, comorbidity, presence of symptoms, type of surgery (emergency or elective), ENETS TNM stage, WHO 2019 grading of the primary tumor, type of resection (R0/1 vs. R2), administration of SSA therapy, duration of follow-up, were collected
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2000-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
re-hospitalization rate for any cause | through study completion, an average of 7 years
  the re-hospitalization rate for any cause after primary tumor surgery

SECONDARY OUTCOMES:
re-hospitalization rate for biliary stone disease | through study completion, an average of 7 years
  the re-hospitalization rate for biliary stone disease after primary tumor surgery
mean number of re-hospitalization any cause | through study completion, an average of 7 years
  the mean number of re-hospitalization for any cause after primary tumor surgery
mean number of re-hospitalization biliary stone disease | through study completion, an average of 7 years
  the mean number of re-hospitalization for biliary stone disease after primary tumor surgery
total costs | through study completion, an average of 7 years
  total costs for primary tumor surgery plus any re-hospitalization
COmplication rate | through study completion, an average of 7 years
  COmplication rate after primary tumor resection

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Ingaldi, MD, Principal Investigator — Azienda Ospedaliero Universitaria, Ospedale S.Orsola Malpighi

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR